CLINICAL TRIAL: NCT04974242
Title: PhysiOtherapist-led Exercise Versus Waiting-list Control for patiEnts Awaiting Rotator Cuff Repair Surgery: a Pilot Randomised Controlled Trial
Brief Title: Physiotherapy for Patients Awaiting Rotator Cuff Repair
Acronym: POWER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospitals of Derby and Burton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UHDB/2021/016
Record Dates: First submitted 2021-06-09; First posted 2021-07-23 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Rotator Cuff Tears
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physiotherapist-led exercise (Experimental): Structured and progressive physiotherapist-led exercise programme. Reflective of current guidance for exercise programmes for people with rotator cuff disorders, an individualised programme developed in relation to the participant's specific goals will be prescribed by the physiotherapist and supported over approximately six contact sessions across a 12-week period.
  Interventions: Other: Physiotherapist-led exercise
- Waiting-list control (No Intervention): Continue on the waiting list for rotator cuff repair surgery, as per usual care.

INTERVENTIONS:
Other: Physiotherapist-led exercise — A programme of physiotherapist-led exercise over approximately 12 weeks.
  Arms: Physiotherapist-led exercise

SUMMARY:
POWER is a pragmatic multi-centre, external pilot randomised controlled trial with feasibility objectives using a parallel group design with 1:1 allocation ratio and integrated qualitative study. The study aims to answer the question: In adult patients diagnosed with tears of the rotator cuff and awaiting elective surgical repair, is it feasible to conduct a future, fully powered, multi-site RCT to test the hypothesis that physiotherapist-led exercise is superior to waiting-list control in terms of clinical and cost-effectiveness?

DETAILED DESCRIPTION:
Tears of the shoulder rotator cuff tendons are a common cause of shoulder pain, disability, and absence from work. Once a decision to undergo rotator cuff repair surgery has been made, patients are placed on a waiting list, and it can take weeks or months to receive the surgery. While waiting for surgery, many patients continue to experience significant pain and disability, and some will be unable to work.

If treatment could be delivered to patients while on the waiting list with potential to reduce pain and disability, and also potentially reduce the need for surgery, there would be clear and significant patient benefit and also benefit to the NHS.

In this pilot study, the investigators will aim to find if it is possible to carry out a larger study to determine if a programme of physiotherapist-led exercise for patients awaiting surgery to repair torn shoulder rotator cuff tendons is clinically and cost-effective.

Working with 4 NHS hospitals, the investigators will recruit 76 patients waiting for rotator cuff repair surgery. One group of patients will receive a programme of specific exercise, supported by a physiotherapist. The second group will just continue waiting for surgery without additional treatment, which is current standard care. The programme of specific exercise can be supported over the telephone, via secure video platform, or face-to-face. the investigators will monitor patients through the study by asking participants to complete one questionnaire at the start and then three more electronic questionnaires after 6 weeks, 3 months and 6 months.

The investigators will invite approximately 25 patients to take part in an interview to discuss experience of the treatments and the study.

The study is being funded by the UK National Institute for Health Research.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients on the elective orthopaedic waiting list for surgical repair of the rotator cuff.

Exclusion Criteria:

* Unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2021-09-29 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Numbers of eligible patients. | 6 months
  Numbers of patients screened and then deemed eligible will be reported descriptively.
Rate of recruitment. | 6 months
  Numbers of patients approached and then randomised as a proportion of the number of eligible patients will be reported descriptively.
Reasons for patients not wanting to participate. | 6 months
  Reasons for patients not wanting to participate will be reported descriptively.
Treatment fidelity (numbers of participants who receive physiotherapy) relating to the programme of physiotherapist-led exercise. | 6 months
  Numbers of participants who receive physiotherapy will be reported descriptively.
Treatment fidelity (number of appointments attended) relating to the programme of physiotherapist-led exercise. | 6 months
  The number of appointments attended will be reported descriptively.
Treatment fidelity (self-report exercise adherence) relating to the programme of physiotherapist-led exercise. | 6 months
  Self-report exercise adherence (intervention group only) will be reported descriptively.
Completion rate of clinical outcome measures. | 6 weeks
  The proportion of clinical outcome questionnaires completed at 6-weeks post-randomisation, including via minimal data collection, will be reported descriptively.
Completion rate of clinical outcome measures. | 3 months
  The proportion of clinical outcome questionnaires completed at three months post-randomisation, including via minimal data collection, will be reported descriptively.
Completion rate of clinical outcome measures. | 6 months
  The proportion of clinical outcome questionnaires completed at six months post-randomisation, including via minimal data collection, will be reported descriptively.
Number and nature of adverse events. | 6 months
  The number and nature of adverse events which occur will be reported descriptively overall and by study arm.
Proportion of participants who report an intention to proceed to surgery or who have received surgery. | 6 months
  The proportion of participants who report an intention to proceed to surgery or who have received surgery within six-months post randomisation will be reported descriptively.

SECONDARY OUTCOMES:
Pain and disability assessed using the Shoulder Pain & Disability Index (SPADI) | 6 weeks, 3 and 6 months post-randomisation
  The SPADI is a 13-item shoulder-specific self-report measure of shoulder pain and disability. The SPADI is reliable, valid, responsive and acceptable to patients. Overall score ranges from 0 to 100, with 0 being the best outcome.
Health related quality of life assessed using the EQ-5D-5L | 6 weeks, 3 and 6 months post-randomisation
  The EQ-5D-5L is a generic measure of health related quality of life that can be used for the purpose of clinical and health economic evaluation. The EQ-5D-5L consists of questions relating to five health domains and respondents rate their degree of impairment using five response levels (no problems, slight problems, moderate problems, severe problems and extreme problems). The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. A total of 3125 possible health states can be defined in this way which can then be converted in to a single index value between 0 and 1, where a higher score indicates a better health state.
Days lost from work due to the shoulder problem | 6 weeks, 3 and 6 months post-randomisation
  Days lost from work due to the shoulder problem will be recorded descriptively on a self-report questionnaire
Days lost from driving | 6 weeks, 3 and 6 months post-randomisation
  Days lost from driving due to the shoulder problem will be recorded descriptively on a self-report questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Chris Littlewood, Study Chair — Manchester Met University
Locations (1):
- University Hospitals Derby and Burton NHS Foundation Trust, Derby, Derbyshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The anonymised datasets generated during and/or analysed during the current study are/will be available upon request from the chief investigator.
  Only de-identified data will be available for request in aggregated format or at the level of the individual participant.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Following publication of the study results and for up to 10 years thereafter.
Access Criteria: An email request should be sent to the chief investigator outlining the type of data to be obtained, the reason for obtaining this data (research question / objective), and the timing for when the data is required to be available (start date/end date). The chief investigator will check that the data set requested is appropriately suited to answer the research question/objective and that the request fits with the original ethical approval and participant consent and adheres to funder and legal restrictions.

DOCUMENTS (1):
  • Study Protocol (2021-06-08): https://cdn.clinicaltrials.gov/large-docs/42/NCT04974242/Prot_000.pdf